CLINICAL TRIAL: NCT02546362
Title: A Single Center, Pilot, Open Trial of the Cefaly® Device in the Treatment of Patients With Fibromyalgia.
Brief Title: Cefaly® Device in the Treatment of Patients With Fibromyalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50212
Record Dates: First submitted 2015-09-09; First posted 2015-09-10 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cefaly active device (Experimental): 12 weeks of treatment using Cefaly twice a day (treatment session of 20 minutes)
  Interventions: Device: Cefaly

INTERVENTIONS:
Device: Cefaly

SUMMARY:
The objective of this pilot open trial was to assess the efficacy and safety of external trigeminal nerve stimulation (e-TNS) with the Cefaly® device in fibromyalgia.

DETAILED DESCRIPTION:
The main objective of this clinical pilot trial was to evaluate the use of external trigeminal nerve stimulation (e-TNS) with the Cefaly® neurostimulator device as a new therapeutic treatment for fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from18 to 65 years (on the day of signing the informed consent form).
2. Diagnosed with fibromyalgia according to the 2010 American College of Rheumatology Preliminary Diagnostic Criteria for Fibromyalgia (ACR 2010).
3. Having a minimum pain score of at least 4 on the 0-10 Fibromyalgia Impact Questionnaire-revised (FIQR) pain scale at screening and baseline.

Exclusion Criteria:

1. Women: Pregnant, lactating or <6 months post partum.
2. Episodic or Chronic Migraine according to the diagnostic criteria listed in International Classification of Headache Disorders (ICHD)-3 beta (2013) section 1, migraine 1, having two or more attacks per month.
3. Change in any medication acting on the central nervous system (CNS) within 28 days before start of the study or during the study.
4. Severe depression i.e. having a Beck Depression Inventory-Fast Screen (BDI-FS) score >12.
5. Botox injection within 4 months before baseline or during the study.
6. Psychiatric disorders that could interfere with study participation: bipolar disorder, psychotic disorders and dementia.
7. Suicidal behavior and/or ideation i.e. having a Columbia Suicide Severity Rating Scale (C-SSRS) score ≥ 4 during the preceding 2 years.
8. Patients currently taking any opioid medication.
9. Patients currently taking medically prescribed marijuana.
10. Current or history during the preceding year of alcohol or substance abuse including marijuana.
11. Widespread rheumatic diseases (other than fibromyalgia), evidence of inflammatory rheumatic disease.
12. Any unstable medical condition in the judgment of the investigator that would interfere with study participation or study assessments.
13. Implanted active metal or electrical devices in the head.
14. Cardiac pacemaker or implanted or wearable defibrillator.
15. Intolerance to supraorbital neurostimulation that makes the treatment not applicable (test of nociceptive threshold with specific Cefaly program).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Arnold, M.D., Principal Investigator — University of Cincinnati; Pierre Rigaux, Study Director — Cefaly Technology
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefaly Active Device: 12 weeks of treatment using Cefaly twice a day (treatment session of 20 minutes
Period: 4-week Treatment Period
Arm/Group | Cefaly Active Device
Started | 50
Completed | 47
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Change in medication | 2
Period: 12-week Treatment Period
Arm/Group | Cefaly Active Device
Started | 47
Completed | 38
Not Completed | 9
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 2
Not completed — Change in medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.10 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Fibromyalgia Impact Questionnaire-revised (FIQR) pain score [Mean (Standard Deviation); unit: score on a scale] — Fibromyalgia Impact Questionnaire-revised (FIQR) pain score is defined on a numeric rating scale scoring the pain between 0 (=no pain) and 10 (=unbearable pain).
  score on a scale | 6.14 (1.29)
Fibromyalgia Impact Questionnaire-revised (FIQR) total score [Mean (Standard Deviation); unit: units on a scale] — Fibromyalgia Impact Questionnaire-revised (FIQR) total score is ranging from 0 to 100, where lower score corresponds to a better quality of life.
  units on a scale | 53.59 (15.32)
EuroQol 5-dimensions - 3-level (EQ-5D-3L) VAS score [Mean (Standard Deviation); unit: units on a scale] — EuroQol 5-dimensions - 3-level (EQ-5D-3L) VAS score is defined on a Visual Analogue Scale (VAS) ranging from 0 (= worth imaginable health state) to 100 (=best imaginable health state).
  units on a scale | 57.49 (17.14)
Patient Reported Outcomes Measurement Information System (PROMIS) score for depression [Mean (Standard Deviation); unit: units on a scale] — Patient Reported Outcomes Measurement Information System (PROMIS) score for depression is ranging from 8 to 40 where higher score is associated with higher depression level.
  units on a scale | 17.06 (5.24)
Patient Reported Outcomes Measurement Information System (PROMIS) score for fatigue [Mean (Standard Deviation); unit: units on a scale] — Patient Reported Outcomes Measurement Information System (PROMIS) score for fatigue is ranging from 8 to 40 where higher score is associated with higher fatigue level.
  units on a scale | 31.12 (4.90)
Patient Reported Outcomes Measurement Information System (PROMIS) score for sleep disturbance [Mean (Standard Deviation); unit: units on a scale] — Patient Reported Outcomes Measurement Information System (PROMIS) score for sleep disturbance is ranging from 8 to 40 where higher score is associated with higher sleep disturbance level.
  units on a scale | 25.86 (5.10)
Multiple Ability Self-report Questionnaire (MASQ) score [Mean (Standard Deviation); unit: units on a scale] — Multiple Ability Self-report Questionnaire (MASQ) score is ranging from 38 to 190, where higher score indicates more difficulty.
  units on a scale | 91.28 (16.04)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity (Fibromyalgia Impact Questionnaire-revised (FIQR) Pain Score) Between Baseline and 12-week Timepoint
Description: Pain intensity (Fibromyalgia Impact Questionnaire-revised (FIQR) pain score) is defined on a numeric rating scale scoring the pain between 0 (=no pain) and 10 (=unbearable pain).
Time Frame: between baseline and 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | -1.33 (2.41)

2. Primary Outcome: Change in Fibromyalgia Impact Questionnaire-revised (FIQR) Total Score Between Baseline and 12-week Timepoint
Description: Fibromyalgia Impact Questionnaire-revised (FIQR) total score is ranging from 0 to 100, where lower score corresponds to a better quality of life.
Time Frame: between baseline and 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | -9.91 (18.51)

3. Secondary Outcome: Change in Pain Intensity (Fibromyalgia Impact Questionnaire-revised (FIQR) Pain Score) Between Baseline and 4-week Timepoint
Description: as for outcome 1
Time Frame: between baseline and 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | -1.45 (2.41)

4. Secondary Outcome: Change in Fibromyalgia Impact Questionnaire-revised (FIQR) Total Score Between Baseline and 4-week Timepoint
Description: as for outcome 2
Time Frame: between baseline and 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | -11.92 (16.18)

5. Secondary Outcome: Patient Global Impression of Change (PGIC) at 4-week Timepoint
Description: Patient Global Impression of Change (PGIC) is defined on a 7-level scale where 1=very much improved and 7=very much worse (4=no change).
Time Frame: at 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | 3.36 (1.11)

6. Secondary Outcome: Patient Global Impression of Change (PGIC) at 12-week Timepoint
Description: as for outcome 5
Time Frame: at 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | 3.33 (1.06)

7. Secondary Outcome: Change in EuroQol 5-dimensions - 3-level (EQ-5D-3L) VAS Score Between Baseline and 4-week Timepoint
Description: EuroQol 5-dimensions - 3-level (EQ-5D-3L) VAS score is defined on a Visual Analogue Scale (VAS) ranging from 0 (= worth imaginable health state) to 100 (=best imaginable health state).
Time Frame: between baseline and 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | 5.79 (15.32)

8. Secondary Outcome: Change in EuroQol 5-dimensions - 3-level (EQ-5D-3L) VAS Score Between Baseline and 12-week Timepoint
Description: as for outcome 7
Time Frame: between baseline and 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | 5.60 (17.05)

9. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Measure for Depression Between Baseline and 4-week Timepoint
Description: Patient Reported Outcomes Measurement Information System (PROMIS) score for depression is ranging from 8 to 40 where higher score is associated with higher depression level.
Time Frame: between baseline and 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | -0.85 (4.47)

10. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Measure for Depression Between Baseline and 12-week Timepoint
Description: as for outcome 9
Time Frame: between baseline and 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | -1.36 (4.95)

11. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Measure for Fatigue Between Baseline and 4-week Timepoint
Description: Patient Reported Outcomes Measurement Information System (PROMIS) score for fatigue is ranging from 8 to 40 where higher score is associated with higher fatigue level.
Time Frame: between baseline and 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | -4.62 (5.35)

12. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Measure for Fatigue Between Baseline and 12-week Timepoint
Description: as for outcome 11
Time Frame: between baseline and 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | -4.00 (6.73)

13. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Measure for Sleep Disturbance Between Baseline and 4-week Timepoint
Description: Patient Reported Outcomes Measurement Information System (PROMIS) score for sleep disturbance is ranging from 8 to 40 where higher score is associated with higher sleep disturbance level.
Time Frame: between baseline and 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | -3.85 (6.36)

14. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Measure for Sleep Disturbance Between Baseline and 12-week Timepoint
Description: as for outcome 13
Time Frame: between baseline and 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | -3.54 (6.35)

15. Secondary Outcome: Change in Multiple Ability Self-report Questionnaire (MASQ) Between Baseline and 4-week Timepoint
Description: Multiple Ability Self-report Questionnaire (MASQ) score is ranging from 38 to 190, where higher score indicates more difficulty.
Time Frame: between baseline and 4-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 47
score on a scale | -2.55 (10.35)

16. Secondary Outcome: Change in Multiple Ability Self-report Questionnaire (MASQ) Between Baseline and 12-week Timepoint
Description: as for outcome 15
Time Frame: between baseline and 12-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cefaly Active Device
Number analyzed (Participants) | 38
score on a scale | -4.74 (13.41)

ADVERSE EVENTS:
Time Frame: The data was collected during the 12 weeks of the treatment period.
Groups:
- Active: 12 weeks of treatment using Cefaly twice a day (treatment session of 20 minutes)
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 40/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=50)
Headache (Nervous system disorders) | 11 (34) — Expected side effect of the Cefaly® device
Nausea (Nervous system disorders) | 2 (2) — Expected side effect of the Cefaly® device
Neck pain (Nervous system disorders) | 3 (4) — Expected side effect of the Cefaly® device
Forehead pain during the session (Nervous system disorders) | 7 (9) — Expected side effect of the Cefaly® device
Persistence of sensation (Nervous system disorders) | 1 (1) — Expected side effect of the Cefaly® device
Sedative effect (Nervous system disorders) | 9 (11) — Expected side effect of the Cefaly® device
Skin reaction (Skin and subcutaneous tissue disorders) | 7 (7) — Expected side effect of the Cefaly® device
Tooth pain (Nervous system disorders) | 2 (2) — Expected side effect of the Cefaly® device
Eye watering, tears (Nervous system disorders) | 2 (2) — Expected side effect of the Cefaly® device
Shingles outbreak (Skin and subcutaneous tissue disorders) | 1 (3) — Unexpected side effect of the Cefaly® device
Worsening fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Unexpected side effect of the Cefaly® device
Dizziness (Nervous system disorders) | 4 (6) — Unexpected side effect of the Cefaly® device
Increase in sinus pain (Nervous system disorders) | 1 (1) — Unexpected side effect of the Cefaly® device
Spacey feeling (Nervous system disorders) | 1 (1) — Unexpected side effect of the Cefaly® device
Normal sensation of the Cefaly® device (Skin and subcutaneous tissue disorders) | 12 (20) — Including itching/tingling/stinging/twitching/vibration/numbness on forehead, scalp, eyes, eyelids, face, lips. But that did not result in treatment permanent discontinuation; these events should have not been considered as Adverse Events.
Burning sensation on forehead or scalp, in eyelids or eyebrows (Skin and subcutaneous tissue disorders) | 2 (7) — Normal sensation of the Cefaly® device but that did not result in treatment permanent discontinuation; these events should have not been considered as Adverse Events
Heaviness in eyelids (Nervous system disorders) | 2 (2) — Normal sensation of the Cefaly® device but that did not result in treatment permanent discontinuation; these events should have not been considered as Adverse Events
Forehead pressure (Nervous system disorders) | 12 (15) — Normal sensation of the Cefaly® device but that did not result in treatment permanent discontinuation; these events should have not been considered as Adverse Events
Headache (Nervous system disorders) | 4 (9) — Relation to the device not suspected
Sinus pressure (Nervous system disorders) | 1 (1) — Relation to the device not suspected
Worsening IBS (Irritable Bowel Syndrome) (Renal and urinary disorders) | 1 (1) — Relation to the device not suspected
Low back spasms (Musculoskeletal and connective tissue disorders) | 1 (1) — Relation to the device not suspected
Flu infection, Cold virus infection, Sinus infection (Infections and infestations) | 4 (5) — Relation to the device not suspected
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Relation to the device not suspected
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) — Relation to the device not suspected
Back pain and stiffness (Nervous system disorders) | 1 (1) — Relation to the device not suspected
Worsening fatigue (Nervous system disorders) | 1 (1) — Relation to the device not suspected
Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 (1) — Relation to the device not suspected
Gastrointestinal virus (Infections and infestations) | 2 (2) — Relation to the device not suspected
Right knee injury (Surgical and medical procedures) | 1 (1) — Relation to the device not suspected
Multiple joint pain (Musculoskeletal and connective tissue disorders) | 1 (2) — Relation to the device not suspected
Back strain (Musculoskeletal and connective tissue disorders) | 2 (2) — Relation to the device not suspected
Tubal ligation (Surgical and medical procedures) | 1 (1) — Relation to the device not suspected
Increase in depression (Psychiatric disorders) | 1 (1) — Relation to the device not suspected
Rash on ankles (Skin and subcutaneous tissue disorders) | 1 (1) — Relation to the device not suspected
Diarrhea (Gastrointestinal disorders) | 2 (2) — Relation to the device not suspected
Vertigo (Nervous system disorders) | 1 (1) — Relation to the device not suspected
Blurred vision (Nervous system disorders) | 1 (1) — Relation to the device not suspected
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Relation to the device not suspected
Viral respiratory illness (Infections and infestations) | 1 (1) — Relation to the device not suspected
Panic attack (Psychiatric disorders) | 1 (1) — Relation to the device not suspected
Restlessness (Nervous system disorders) | 2 (2) — Relation to the device not suspected
Worsening right knee or foot pain (Nervous system disorders) | 2 (2) — Relation to the device not suspected
Swollen right thigh and knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Relation to the device not suspected
Ringing in the ears/Ears ache (Ear and labyrinth disorders) | 3 (3) — Relation to the device not suspected
Burning sensation in both legs and right shoulder (Skin and subcutaneous tissue disorders) | 1 (1) — Relation to the device not suspected
Body tingling (Skin and subcutaneous tissue disorders) | 1 (1) — Relation to the device not suspected
Cold sensation in left cheek (Nervous system disorders) | 1 (3) — Relation to the device not suspected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 45 days from the time submitted to the sponsor for review. Sponsor may request:

* deletion of any trade secret, proprietary, or confidential information of Sponsor
* an additional 60 days to take measures to preserve its Intellectual Property rights

Sponsor's written consent is required for results communication before trial completion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT02546362/Prot_SAP_000.pdf